CLINICAL TRIAL: NCT04183504
Title: Early STEPs: Screening for Therapy and Empowering Parents: A Pilot Study
Brief Title: Screening for Therapy and Empowering Parents: A Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Tennessee (Other)
Responsible Party: Principal Investigator, Anne Zachry, Chair, Department of Occupational Therapy, Principle Investigator, Associate Professor, University of Tennessee
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 14-03212-XP
Record Dates: First submitted 2019-11-25; First posted 2019-12-03 (Actual); Last update posted 2023-05-18 (Actual); Status verified 2023-05

CONDITIONS: Primary Health Care
Keywords: Primary Health Care; Occupational Therapy; Child Development; Early Intervention; Parenting

STUDY DESIGN:
Intervention Model Description: One group pretest-posttest design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Early Steps Coaching (Experimental): Coaching session on positive parenting practices and promoting child development.
  Interventions: Behavioral: Brief parenting intervention

INTERVENTIONS:
Behavioral: Brief parenting intervention — Coaching session on positive parenting practices and promoting child development

SUMMARY:
The purpose of this study is expand on the Early STEPs project goal of identifying early developmental delays in infants and young children in a health disparate population and to collect preliminary data to lay the groundwork for a future NIH grant proposal. Individuals with less education have poor health and shorter life expectancies than well-educated individuals, and research reveals that poverty is directly related to limited education. An innovative approach is needed to overcome barriers, improve health literacy, and educate parents on effective parenting strategies for this population. Technology may be the part of the solution to this issue. Through Early STEPs, the occupational therapists will continue to refer families to early intervention and therapy services as appropriate and follow-up to ensure that services are initiated. The Occupational Therapist will also determine if the parents are utilizing the Word Gap App and other provided resources to support their child's development and to manage their stress. By increasing parental awareness and knowledge of language and motor skill development, the environments of underserved children will be enriched and parental stress will be reduced so that these children can have improved health and reach their full potential.

DETAILED DESCRIPTION:
1. Purpose: The purpose of this study is to determine the effectiveness of developmental screening to identify developmental delays in order to make appropriate referrals for early intervention services.
2. Rationale: Research has consistently shown that providing timely early intervention (EI) services for young children identified as developmentally delayed improves both short-term and long-term outcomes. It is critical that children with delays be identified as early as possible because intervention programs are more effective when initiated at a young age. In fact, the American Academy of Pediatrics (AAP) advocates identifying delays before children reach 2 years of age.

   There is evidence that primary care providers tend to under-detect developmental delays among infants and young children. In addition, in high poverty areas, transportation, finances and other logistical challenges often prevent parents of young children from regularly visiting a physician, which further contributes to limited opportunities for intervention.

   Under-enrollment in intervention programs has been identified as a national problem, one that is recognized as a critical issue in the Mid-South due to the lower percentage of young children being identified and referred for services. Nationally, it is estimated that 16-18% of children have disabilities; however, less than one-third of these cases are referred for intervention before kindergarten age. Besides the issue of under-identification of developmental problems in young children, research suggests that many children who are referred for Early Intervention services do not end up receiving therapy due to poor follow-through by caregivers. It is likely that families need support and guidance regarding the importance of Early Intervention services.

   Unaddressed developmental delays can negatively impact the future health and educational attainment of our nation's infants. Families benefit from screening through an increased awareness of appropriate developmental and behavioral expectations. For example, screening can lead to positive outcomes in family interaction and decreased parental stress levels when developmental information and recommendations for activities are provided, even for children who do not fully meet the criteria to be referred. In the Memphis area, enrollment of children under the age of 3 in EI programs has actually decreased over the past five years, despite strong evidence that the incidence of disabilities such as autism is on the rise. Nationally, 2.52% of young children receive EI services; in Tennessee, 1.8% of children are receiving services needed.
3. Study/Project Population: Through the Early STEPs Project, licensed occupational therapists will provide free developmental and autism screenings to children ages birth to and 6 years 11 months 29 days in a pediatric medical practice.
4. Research Design: To determine the effectiveness of the Early STEPs project, investigators will compare pre- and post-project referrals for EI services, follow through by families, and pre and post parental satisfaction qualitative data. The participating pediatric practices will provide documentation of their prior average number of monthly early intervention referrals and this information will be compared to the monthly number of referrals at the end of the study period. The investigators will follow-up with the parent of the referred child at 6- and 12-months to determine if early intervention services were initiated by the parent and to determine if the parents perceived that the developmental app and online support group were helpful and improved confidence with their parenting skills.

   The data collection will begin on February 3, 2014 and end in approximately 2 years.
5. Procedures The developmental screenings will be offered two to four days per month. Informational flyers will be posted locally and in the pediatrician's offices. Investigators will obtain parental consent. If parental consent is obtained, the screenings will be conducted with the parent present. The process will involve the parents providing qualitative information regarding the confidence with their parenting skills, and the occupational therapy investigators will complete The Ages & Stages Questionnaire (ASQ-3) on each participant and the Modified Checklist for Autism in Toddlers, if age appropriate to the particular child. All information for the screenings will be collected from the parent. Researchers will not be accessing the subjects' medical records. Additionally, early intervention/parental coaching sessions will be provided by occupational therapists as needed. Caregivers will utilize skills training, free online resources and an online social support network to develop and maintain nurturing parenting skills. Follow-up phone calls will take place at 6-months and 12-months after a positive screening to determine if therapy services were indicated and to determine if the use of online resources or the social support network were perceived to be helpful. During the 6 and 12-month follow-up phone call, study personnel will collect information regarding parenting confidence using the Parenting Sense of Competence Scale (PSCO). Parents or caregivers will receive a free t-shirt as available and a developmental flyer for participating. (Courtesy of The Urban Child Institute). Parents or caregivers will receive free first year milestone applications for their cellular devices (courtesy of Aimee's Babies).
6. Outcome Measures: The PI will monitor and report on:

   1. number of children identified for further assessment,
   2. common developmental concerns/delays,
   3. specific services referred to,
   4. Caregiver follow-up
   5. The investigators will collect data using the PSCO regarding parenting confidence at the initial visit and during the 6 and 12-month follow-up phone call.

ELIGIBILITY:
Inclusion Criteria:

* parent provides written informed consent to take part in the study
* child has no congenital malformations or genetic syndromes
* child is not enrolled in Early Intervention Services.
* child is not in foster care
* Parent agrees to attend parent training session
* Parent agrees to complete pre- and post- Parenting Sense of Competence scale
* Child is between birth and 6 years 11 months 29 days

Exclusion Criteria

* Parent will not signed informed consent.
* child has congenital malformations or genetic syndrome
* child is not enrolled in Early Intervention Services.
* child is in foster care
* child is 7 years or older

Max Age: 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2015-11-01 (Actual); Primary Completion 2018-05-07 (Actual); Study Completion 2018-05-07 (Actual)

PRIMARY OUTCOMES:
Parenting Sense of Competence Scale | Through study completion, an average of 2 years.
  Parenting Sense of Competence Scale- Scores range from 9 to 54, with higher scores indicating greater parenting satisfaction.

SECONDARY OUTCOMES:
Developmental screening results | Through study completion, an average of 2 years.
  Ages & Stages Questionniare03 (ASQ-3TM), parental report questionnaire that provides scores for each of the following domains: communication, gross motor, fine motor, problem- solving, and personal/social skills. Every version of the screening includes specific cutoff scores to indicate if child's development is on schedule or not. The cutoff scores vary from one age level to the next, ranging from 0 to 60, with 60 indicating a higher developmental level.
Number of referrals for early intervention or therapy services | Through study completion, an average of 2 years.
  Actual number of referrals made to early intervention services or therapy.
Follow through in obtaining early intervention or therapy services | Through study completion, an average of 2 years.
  Counts for each type of service obtained: early intervention, occupational therapy, physical therapy, speech therapy, or comprehensive developmental evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Anne H Zachry, PhD, Principal Investigator — University of Tennessee
Locations (2):
- United States (2):
  - Memphis Children's Clinic, Memphis, Tennessee
  - University of Tennessee Health Science Center, Memphis, Tennessee

IPD SHARING:
Plan to Share IPD: Yes
Study protocol, Statistical Analysis Plan, Informed Consent Form
Supporting Information: Study Protocol, SAP
Time Frame: Immediately
Access Criteria: Contact PI @ azachry@uthsc.edu

REFERENCES:
- [Result] Berry AD, Garzon DL, Mack P, Kanwischer KZ, Beck DG. Implementing an early childhood developmental screening and surveillance program in primary care settings: lessons learned from a project in Illinois. J Pediatr Health Care. 2014 Nov-Dec;28(6):516-25. doi: 10.1016/j.pedhc.2014.04.008. Epub 2014 Jun 11. PMID 24929846
- [Result] Council on Children With Disabilities; Section on Developmental Behavioral Pediatrics; Bright Futures Steering Committee; Medical Home Initiatives for Children With Special Needs Project Advisory Committee. Identifying infants and young children with developmental disorders in the medical home: an algorithm for developmental surveillance and screening. Pediatrics. 2006 Jul;118(1):405-20. doi: 10.1542/peds.2006-1231. PMID 16818591
- [Result] Dobrez D, Sasso AL, Holl J, Shalowitz M, Leon S, Budetti P. Estimating the cost of developmental and behavioral screening of preschool children in general pediatric practice. Pediatrics. 2001 Oct;108(4):913-22. doi: 10.1542/peds.108.4.913. PMID 11581444
- [Result] Earls MF, Hay SS. Setting the stage for success: implementation of developmental and behavioral screening and surveillance in primary care practice--the North Carolina Assuring Better Child Health and Development (ABCD) Project. Pediatrics. 2006 Jul;118(1):e183-8. doi: 10.1542/peds.2006-0475. PMID 16818532
- [Result] Frankenburg WK. Developmental surveillance and screening of infants and young children. Pediatrics. 2002 Jan;109(1):144-5. doi: 10.1542/peds.109.1.144. No abstract available. PMID 11773555
- [Result] Guevara JP, Gerdes M, Localio R, Huang YV, Pinto-Martin J, Minkovitz CS, Hsu D, Kyriakou L, Baglivo S, Kavanagh J, Pati S. Effectiveness of developmental screening in an urban setting. Pediatrics. 2013 Jan;131(1):30-7. doi: 10.1542/peds.2012-0765. Epub 2012 Dec 17. PMID 23248223
- [Result] Rosenberg SA, Zhang D, Robinson CC. Prevalence of developmental delays and participation in early intervention services for young children. Pediatrics. 2008 Jun;121(6):e1503-9. doi: 10.1542/peds.2007-1680. Epub 2008 May 26. PMID 18504295
- [Result] Rydz D, Srour M, Oskoui M, Marget N, Shiller M, Birnbaum R, Majnemer A, Shevell MI. Screening for developmental delay in the setting of a community pediatric clinic: a prospective assessment of parent-report questionnaires. Pediatrics. 2006 Oct;118(4):e1178-86. doi: 10.1542/peds.2006-0466. PMID 17015506
- [Result] Schonwald A, Huntington N, Chan E, Risko W, Bridgemohan C. Routine developmental screening implemented in urban primary care settings: more evidence of feasibility and effectiveness. Pediatrics. 2009 Feb;123(2):660-8. doi: 10.1542/peds.2007-2798. PMID 19171635